CLINICAL TRIAL: NCT04374539
Title: Plasma Exchange in Patients With COVID-19 Disease and Invasive Mechanical Ventilation: a Randomized Controlled Trial
Acronym: REP-COVID
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: inability to recruit more patients
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Project Manager, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-001722-66
Record Dates: First submitted 2020-05-02; First posted 2020-05-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections | interventions — Plasma Exchange

STUDY DESIGN:
Intervention Model Description: Multicenter open label randomized controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plasma exchange (Experimental): Plasma exchange with human serum albumin + Polyclonal immunoglobulin + standard medical treatment
  Interventions: Biological: Plasma exchange
- Standar medical treatment (Active Comparator): Standar medical treatment
  Interventions: Drug: Standar medical treatmen

INTERVENTIONS:
Biological: Plasma exchange — Plasma exchanges with 5% human albumin and fresh frozen plasma in patients with quick <50% or only with 5% albumin in patients with quick of 50% or more. We will exchange between 1.2 and 1.5 plasma volumes, that will vary according to sex, weight, height and hematocrit.
  Polyclonal immunoglobulin will be administered at a dose of 100 mg / kg ev after each plasma exchange.
  Standar Medical treatment Kaletra:
  lopinavir/ritonavir: 2c/12h 7 days
  * Hydroxychloroquine sulfate 400 mg/12h the first day followed by 200 mg /12h 4 days
  * Azithromycin 500 mg first day, followed by 250 mg /d 4 days (oral or EV)
  * Tocilizumab 400 mg (weight <75Kgs) or 600 mg (weight ≥ 75 Kg)
  * Methylprednisolone 250 mg EV three days and 30 mg/d another 3 days
  * Anakinra 200mg/ 12h SBC first day, 200mg / 24h SBC two more days
  * Clexane 40-60 mg/d
  Arms: Plasma exchange
Drug: Standar medical treatmen — Kaletra: lopinavir/ritonavir: 2c/12h 7 days
  * Hydroxychloroquine sulfate 400 mg/12h the first day followed by 200 mg /12h 4 days
  * Azithromycin 500 mg first day, followed by 250 mg /d 4 days (oral or EV)
  * Tocilizumab 400 mg (weight <75Kgs) or 600 mg (weight ≥ 75 Kg)
  * Methylprednisolone 250 mg EV three days and 30 mg/d another 3 days
  * Anakinra 200mg/ 12h SBC first day, 200mg / 24h SBC two more days
  * Clexane 40-60 mg/d
  Arms: Standar medical treatment

SUMMARY:
Plasma exchanges with 5% human albumin (2/3 of the exchanged plasma volume) and fresh frozen plasma (FFP: 1/3) in patients with quick <50% or only with 5% albumin in patients with quick of 50% or more. We will exchange between 1.2 and 1.5 plasma volumes, that will vary according to sex, weight, height and hematocrit.

DETAILED DESCRIPTION:
Plasma exchange (PE) is a standardized and safe therapeutic procedure, used in the treatment of various diseases that require rapid and prolonged elimination of endogenous and exogenous substances, with deleterious effects on the function of different organs and systems. The efficacy and safety of PE has been demonstrated in patients with fulminant hepatitis (FH), an entity characterized by an exacerbated inflammatory response, multi-organ failure, and high short-term mortality. In FH, plasma exchange improves systemic inflammation, prevents organ failure and renal support requirements, and improves survival. Such treatment eliminates important endogenous and exogenous inducers of the systemic inflammatory response (PAMPs and DAMPs), proinflammatory mediators (cytokines and ROS), and other biologically active substances (nitric oxide, prostaglandins, and bradykinin) that are involved in the pathogenesis of organ failure. Several case reports also suggest that PE is an effective rescue therapy in critically ill patients with influenza A (H1N1). However, the efficacy of PE has not been evaluated in critically ill patients with COVID-19 disease.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject ≥18 years and < 80 years of age;
2. Subjects with diagnosis of COVID-19 disease by PCR in nasopharyngeal smear, sputum, or bronchial aspirates;
3. Subjects admitted in ICU with invasive mechanical ventilation;
4. Informed consent granted via telephone by relatives or legal representative

Exclusion Criteria:

1. More than seven days with invasive mechanical ventilation
2. Refractory Shock (Noradrenaline dose > 0.5 micrograms/ kg/minute)
3. Decompensated Cirrhosis
4. Chronic kidney disease requiring hemodialysis
5. Active neoplastic disease
6. Severe chronic heart failure (NYHA class III or IV)
7. Severe pulmonary disease (GOLD III or IV)
8. HIV infection (AIDS criteria)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-04-29 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2021-06-29 (Actual)

PRIMARY OUTCOMES:
Impact of plasma exchange | 28 days
  Number of exitus at 28 days after plasma exchange in patients with COVID-19 disease and invasive mechanical ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No